CLINICAL TRIAL: NCT04135586
Title: Effects of a Physical Exercise Intervention at the Molecular Systemic and Tumor Level Performed During Neoadjuvant Chemotherapy in Women With Breast Cancer
Brief Title: Effects of a Physical Exercise Intervention During Neoadjuvant Chemotherapy in Women With Breast Cancer
Acronym: NEOLIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Alejandro Lucia, Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UEM Quirón
Record Dates: First submitted 2019-10-08; First posted 2019-10-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Physical Exercise
Keywords: exercise; high interval training; resistance exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Physical exercise intervention (24 weeks)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The patients in this arm will follow an exercise program for 24 weeks (i.e., during neo-adjuvant treatment), with two sessions per week including both aerobic and resistance training. Exercise intensity will range between 65% and 100% of the maximum score in the scale of Rated Perceived Exertion (RPE).
  Interventions: Other: Exercise training
- Control (Other): The patients follow their usual habits as well as a Yoga program. They will also receive educational sessions on the benefits of regular physical activity (brisk walking).
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise training — Exercise program for 24 weeks (with neo-adjuvant treatment), with two sessions per week including both moderate-to-intense aerobic and resistance training. The intensity of each type of exercise will range between 65% and 100% of the maximum score in the Rated Perceived Exertion (RPE) scale.
  Arms: Exercise
Other: Control — Yoga + educational program
  Arms: Control

SUMMARY:
To assess in women with triple-negative breast cancer receiving neo-adjuvant chemotherapy the effects of an intense physical exercise program (intervention group) on physical capacity, compared with a control group not meeting the minimum exercise recommendations of the World Health Organization (WHO).

DETAILED DESCRIPTION:
Justification and aims Breast cancer is the fourth most common type of cancer worldwide and the first among women in Spain. It is also the type of cancer with the highest mortality. Several studies have assessed the effects of exercise performed in the neo-adjuvant period, but there is heterogeneity among them.

Principal aim:

To assess in women with triple-negative breast cancer receiving neo-adjuvant chemotherapy the effects of an intense physical exercise program (intervention group) on physical capacity, compared with a control group not meeting the minimum exercise recommendations of the World Health Organization (WHO).

Secondary aims:

To compare the following outcomes in both groups: body composition, and quality of life and depression/anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast carcinoma in the 'Hospital Universitario Quirónsalud de Pozuelo' (Madrid, Spain) and following neoadjuvant therapy in the aforementioned center.
* Must have triple negative breast cancer (i.e., negative for estrogen receptors, progesterone receptors, and excess HER2 protein) of size > or equal to 15 mm

Exclusion Criteria:

* Not meeting all of the above.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Change from baseline to end of intervention (i.e., after 24 weeks)
  peak rate of oxygen consumption (ml/kg/min) reached during a graded treadmill exercise test until exhaustion
muscle dynamic strength | Change from baseline to end of intervention (i.e., after 24 weeks)
  Time (seconds) to perform the sit-to-stand (STS) test (five consecutive repetitions of sitting down and uprising from a chair)
handgrip strength | Change from baseline to end of intervention (i.e., after 24 weeks)
  handgrip strength measured using a dynamometer and scores recorded in kilograms (to the nearest 0.1 kg)

SECONDARY OUTCOMES:
Health-related quality of life (Breast Cancer-Specific Quality of Life Questionnaire [QLQ-BR23]) | Change from baseline to end of intervention (i.e., after 24 weeks)
  The QLQ-C30 is a multidimensional cancer HRQoL questionnaire that contains 30 items assessing six functional and nine symptom scales. Results from this questionnaire are transformed into scores ranging from 0 to 100 according to European Organization for Research and Treatment of Cancer (EORTC) scoring, with higher scores in the functioning scales indicating a better functional status and global HRQoL, and higher scores on the symptoms' scales indicating more symptoms.
Body composition (fat mass) | Change from baseline to end of intervention (i.e., after 24 weeks)
  fat mass (% of whole body mass), evaluated by dual energy X-ray absorptiometry
Body composition (lean body mass) | Change from baseline to end of intervention (i.e., after 24 weeks)
  lean body mass (% of whole body mass), evaluated by dual energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Quirónsalud de Pozuelo (HUQP), Madrid
  - Lgcortijo@Gmail.Com, Madrid